CLINICAL TRIAL: NCT00986596
Title: A Pilot Study of the Impact of Vitamin D3 on Muscle Performance in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Director, Bone Metabolism Laboratory, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2450; 7528
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Sarcopenia; Falls
Keywords: vitamin D; skeletal muscle; vitamin D receptor
MeSH Terms: conditions — Sarcopenia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D3 (Active Comparator): vitamin D3 capsule 4000 IU p.o. daily
  Interventions: Dietary Supplement: vitamin D3
- placebo (Placebo Comparator): microcrystalline cellulose capsule p.o. daily (identical to vitamin D capsule)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 4000 IU once daily by mouth for 4 months
  Arms: vitamin D3
Dietary Supplement: Placebo — microcrystalline cellulose capsule p.o. daily (identical to vitamin D capsule)
  Arms: placebo

SUMMARY:
The purpose of the study is to investigate the effect of vitamin D on muscle tissue and physical performance.

DETAILED DESCRIPTION:
The investigators have recently observed that among healthy women age 65 and older who participated in a placebo-controlled vitamin D and calcium intervention trial, those treated with supplements had a lower risk of falling than those in the placebo group. Vitamin D receptors (VDRs) are present in muscle tissue and are thought to mediate the favorable effects of vitamin D on muscle performance. Vitamin D insufficiency is common particularly in the elderly and supplementation with a relatively high dose of vitamin D may be a useful approach for improving muscle performance and potentially lowering the risk of falling in sedentary older women and other high-risk populations.

The investigators will aim to study women, age 65 and older, with 25(OH)D levels below 60 nmol/l in a double-blind, 4-month randomized controlled pilot study. Eligible subjects will be randomized to treatment with 4000 IU per day of vitamin D3 or placebo. Blood and 24 hour urine will be measured at the beginning and end of the study as outlined in the intervention and measurement schedule below. In addition, a safety random spot urine will be analyzed for calcium and creatinine on day 30. Muscle performance measures will be measured and muscle biopsies will be performed at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* 25 (OH)D levels >22.5 nmol/l or <60 nmol/l
* Women must have a composite physical performance score of ≤ 9 out of a possible score of 12.
* Subjects must agree not to change their usual level of physical activity or change the amount of calcium and vitamin D supplement they use for the duration of the study.
* If they are taking calcium supplements, they must agree to take the supplement any time after lunch.

Exclusion Criteria:

* General:

  1. Total calcium intake >1000mg daily on the prescreening questionnaire.
  2. More than 400 IU daily of supplemental vitamin D on the prescreening questionnaire.
  3. A screening 25(OH)D level > 60 nmol/ L.
  4. Screening 24-hour urine calcium > 275 mg.
  5. An abnormal serum calcium.
  6. Travel to latitude <35 degrees N within 2 months of the time of enrollment; plans to travel to latitude <35 degrees N during the 4-month study, with the likelihood of tanning (e.g. appreciable sun exposure without sun screen).
  7. Greater than 2 drinks of alcohol a day.
* Medications:

  1. Bone active drugs such as bisphosphonates, estrogen, calcitonin, teriparatide
  2. Diuretics
  3. Oral glucocorticoids in the last month
  4. Phosphates in the last week
  5. Lithium
  6. Cod liver oil
  7. Total parenteral nutrition
  8. Calcium containing antacids
  9. Coumadin or other prescribed anticoagulants
* Diseases:

  1. Active thyroid disease - unstable levothyroxine dose
  2. Parathyroid disease
  3. Sarcoidosis
  4. Fracture of the foot, leg, or hip in the last year
  5. Renal stone < 5 years
  6. Alkaline phosphatase > 10% above the upper limit of normal
  7. Pancreatitis
  8. Active malignancy (other than basal cell cancer of the skin) or cancer therapy in the last year
  9. Uncontrolled arrhythmia in last year
  10. Malabsorption
  11. Use of a walker or wheelchair (3-post cane okay)
  12. Nasal oxygen use
  13. Must have a basic mobility level of walking 4 meters
  14. Hemiplegia
  15. Tuberculosis
  16. Type 1 Diabetes mellitus or unstable type 2 diabetes mellitus (fasting blood glucose >130 mg/dL)
  17. Other abnormality in screening labs, at the discretion of the study physician

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Define and compare changes in size and number of type II muscle fibers in response to 4 months of treatment with 4000 IU of vitamin D3 per day or placebo in older women with low-normal 25(OH)D levels. | 4 months

SECONDARY OUTCOMES:
Define and compare vitamin D signaling in muscle biopsy specimens taken before and after the treatment. | 4 months
Define and compare changes in clinical measures of muscle performance before and after treatment | 4 months
Define and compare levels of bone turnover before and after treatment | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts University; Lisa Ceglia, MD, Study Director — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States